CLINICAL TRIAL: NCT04231474
Title: Urodynamic Evaluation Neurgenic Bladder in Patients After Spinal Cord Injury
Brief Title: Urodynamic Evaluation in Patients After Spinal Cord Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ewa Chlebus, lek.Ewa Chlebuś, Department of Rehabilitation and Physiotherapy Rehabilitation, Poznan University of Medical Sciences
Other Study IDs: 1/2019CReh; 111/19 (Other: Bioethics Committee by the Poznan)
Record Dates: First submitted 2019-11-25; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Spinal Cord Injuries; Neurogenic Bladder; Urodynamics
Keywords: Urodynamics
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Bladder, Neurogenic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Demographic and clinical features of the patients: Number of patients Time from injury to hospitalization Time from injury to urodynamic evaluation Duration of hospitalization
  Interventions: Device: Urodynamic testing
- Comparison of urodynamic outcomes: Treatment options in patients with level SCI : cervical, thoracical and lumbar spinal cord injury
  Interventions: Device: Urodynamic testing

INTERVENTIONS:
Device: Urodynamic testing — All data were obtained using the MMS Alfa 4T by the same urologist with use of an 8 Charr catheter.

SUMMARY:
Retrospective study, which analyzed 100 medical histories of patients who were admitted o the Neurological Rehabilitation Ward of the Rehabilitation Clinic in the Orthopedic-Rehabilitation Hospital in Poznan in years 2010-2019.

DETAILED DESCRIPTION:
All patients considered for the study underwent routine testing: blood counts, urinalysis, urine culture, and sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* incomplete spinal cord injuries,
* the results of the urodynamic testing (conducted by the same urologist) by admission,
* urine culture test by admission.

Exclusion Criteria:

* complete spinal cord injury
* without urodynamic test in medical documentation by admission,
* without urine culture test by admission,
* with symptomatic urinary tract infection in urodynamic test

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Eventually, 54 patients were enrolled in the study (12 women, 42 men). The incompleteness and level of SCI were diagnosed based on MRI, which was performed directly after the injury in Neurosurgery Ward or Trauma Center.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2020-01-20 (Estimated); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Urethra sensation | 30 days after spinal injury,
  2 - preserved, 1- reduced, 0 - absent
Urethra sensation | after 3 months of rehabilitation
  2 - preserved, 1- reduced, 0 - absent
Intravesical pressure | 30 days after spinal injury,
  0- normal, 1- low
Intravesical pressure | after 3 months of rehabilitation
  0- normal, 1- low
Bladder complaince | 30 days after spinal injury,
  2- high, 1- reduced
Bladder complaince | after 3 months of rehabilitation
  2- high, 1- reduced
Bladder stability | 30 days after spinal injury,
  0 -stable, 1- hyperactive
Bladder stability | after 3 months of rehabilitation
  0 -stable, 1- hyperactive
Bladder sensation | 30 days after spinal injury
  2-preserved,1- reduced, 0- absent
Bladder sensation | after 3 months of rehabilitation
  2-preserved,1- reduced, 0- absent
Bladder capacity | 30 days after spinal injury
  ml ( Average, Median, SD)
Bladder capacity | after 3 months of rehabilitation
  ml ( Average, Median, SD)
Urine volume | 30 days after spinal injury
  ml ( Average, Median,SD)
Urine volume | after 3 months of rehabilitation
  ml ( Average, Median,SD)

CONTACTS AND LOCATIONS:
Overall Officials: Przemysław Lisiński, MPhD, Study Director — Clinic Rehabilitation, University of Medical Sciences in Poznań
Locations (1):
- Department of Rehabilitation and Physiotherapy Rehabilitation,, Poznan, Poland

IPD SHARING:
Plan to Share IPD: Undecided
Urodynamic evaluation in patients after spinal cord injury